CLINICAL TRIAL: NCT01498250
Title: Microarray Analysis of microRNA Expression in Basal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Principal Investigator, Ruhr University of Bochum
Other Study IDs: microRNA6
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — basal cell carcinoma and non-lesional skin
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- basal cell carcinoma
- non-lesional skin

SUMMARY:
Perturbations in microRNA (miRNA) expression profiles has been reported for a variety of cancers. This study will be an exploratory analysis of miRNA expression in basal cell carcinoma by miRNA expression profiling using microarrays.

DETAILED DESCRIPTION:
Perturbations in the expression profiles of microRNAs (miRNAs) have been reported for a variety of different cancers. Basal cell carcinoma (BCC) of the skin has not been systematically evaluated regarding differentially expressed miRNAs. Patients with BCC are included in the study to perform an exploratory analysis by miRNA expression profiling using microarrays. Expression levels of miRNA candidates will be validated by TaqMan real-time quantitative polymerase chain reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* Basal Cell Carcinoma

Exclusion Criteria:

* Other Skin Cancer than Basal Cell Carcinoma

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with
  Basal Cell Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Falk G Bechara, PD Dr., Study Director — Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum; Peter Altmeyer, Prof. Dr., Study Chair — Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum; Michael Sand, Dr., Principal Investigator — Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum
Locations (1):
- Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Sand M, Skrygan M, Sand D, Georgas D, Hahn SA, Gambichler T, Altmeyer P, Bechara FG. Expression of microRNAs in basal cell carcinoma. Br J Dermatol. 2012 Oct;167(4):847-55. doi: 10.1111/j.1365-2133.2012.11022.x. Epub 2012 Aug 20. PMID 22540308